CLINICAL TRIAL: NCT03830866
Title: A Phase III, Randomized, Multi-Center, Double-Blind, Global Study to Determine the Efficacy and Safety of Durvalumab in Combination With and Following Chemoradiotherapy Compared to Chemoradiotherapy Alone for Treatment in Women With Locally Advanced Cervical Cancer
Brief Title: Study of Durvalumab With Chemoradiotherapy for Women With Locally Advanced Cervical Cancer (CALLA)
Acronym: CALLA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9100C00001; 2018-002872-42 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2019-02-05 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Durvalumab; Chemoradiotherapy; Locally Advanced Cervical Cancer
MeSH Terms: interventions — durvalumab; Cisplatin; Carboplatin; Brachytherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab (intravenous infusion) (Experimental): durvalumab + standard of care concurrent chemoradiation therapy(SoC CCRT) followed by durvalumab monotherapy up to 24 months or until PD from the date of randomization
  Interventions: Biological: Durvalumab; Drug: Cisplatin; Drug: Carboplatin; Radiation: external beam radiation therapy (EBRT) + brachytherapy
- Placebo (matching placebo for intravenous infusion) (Placebo Comparator): placebo + standard of care concurrent chemoradiation therapy(SoC CCRT)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Radiation: external beam radiation therapy (EBRT) + brachytherapy

INTERVENTIONS:
Biological: Durvalumab — IV infusion every 4 weeks
  Arms: Durvalumab (intravenous infusion)
Drug: Cisplatin — Platinum based Standard of Care Chemotherapy administered concurrent with radiation therapy
Drug: Carboplatin — For patients enrolled under CSP v2 and prior - platinum based Standard of Care Chemotherapy administered concurrent with radiation therapy
Radiation: external beam radiation therapy (EBRT) + brachytherapy — Radiation therapy per standard of care

SUMMARY:
This is a randomized, multi-center, double-blind, placebo-controlled, global, Phase III study to determine the efficacy and safety of durvalumab + Chemoradiotherapy versus Chemoradiotherapy alone as treatment in Women With Locally Advanced Cervical Cancer

DETAILED DESCRIPTION:
Women will be randomized in a 1:1 ratio to receive treatment with concurrent durvalumab + standard of care (SoC) or Placebo + Soc, followed by durvalumab/placebo maintenance for 24 months.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Female
2. Aged at least 18 years
3. Documented evidence of cervical adenocarcinoma or squamous carcinoma FIGO (2009) Stages IB2 to IIB node positive or FIGO (2009) IIIA-IVA any node
4. No prior chemotherapy or radiotherapy for cervical cancer
5. WHO/ECOG performance status of 0-1
6. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 Target Lesion at baseline.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Diagnosis of small cell (neuroendocrine) histology or mucinous adenocarcinoma cervical cancer
2. Intent to administer a fertility-sparing treatment regimen
3. Undergone a previous hysterectomy
4. Evidence of metastatic disease per RECIST 1.1 including lymph nodes ≥15 mm (short axis) above the L1 cephalad body, in the inguinal region or outside the planned radiation field.
5. History of allogeneic organ transplantation
6. Active or prior documented autoimmune or inflammatory disorders
7. Uncontrolled intercurrent illness
8. History of another primary malignancy and active primary immunodeficiency

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female: only female participants are being studied
Enrollment: 770 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urban Scheuring, M.D., Ph.D., Study Director — AstraZeneca; Bradley Monk, M.D, Principal Investigator — University of Arizona, Arizona, USA
Locations (90):
- United States (13):
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Orange, California
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lake Success, New York
  - Research Site, The Bronx, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Spring, Texas
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Fortaleza
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Chile (4):
  - Research Site, Antofagasta
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (11):
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Szeged
- India (8):
  - Research Site, Ahmedabad
  - Research Site, Gūrgaon
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Visakhapatnam
- Japan (11):
  - Research Site, Fukuoka
  - Research Site, Kagoshima
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Nakagami-gun
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Toon-shi
  - Research Site, Yokohama
- Mexico (7):
  - Research Site, Alc. Cuauhtémoc
  - Research Site, Deleg. Tlalpan
  - Research Site, Guadalajara
  - Research Site, Guadalajara Jalisco
  - Research Site, Mérida
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
- Research Site, Lima, Peru
- Philippines (6):
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Iloilo City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Lodz
  - Research Site, Lublin
- Russia (5):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Kaluga
  - Research Site, Moscow
  - Research Site, Novosibirsk
- South Africa (2):
  - Research Site, Parktown
  - Research Site, Port Elizabeth
- Research Site, Seoul, South Korea
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Monk BJ, Toita T, Wu X, Vazquez Limon JC, Tarnawski R, Mandai M, Shapira-Frommer R, Mahantshetty U, Del Pilar Estevez-Diz M, Zhou Q, Limaye S, Godinez FJR, Oppermann Kussler C, Varga S, Valdiviezo N, Aoki D, Leiva M, Lee JY, Sulay R, Kreynina Y, Cheng WF, Rey F, Rong Y, Ke G, Wildsmith S, Lloyd A, Dry H, Tablante Nunes A, Mayadev J. Durvalumab versus placebo with chemoradiotherapy for locally advanced cervical cancer (CALLA): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Dec;24(12):1334-1348. doi: 10.1016/S1470-2045(23)00479-5. PMID 38039991
- [Derived] Mayadev J, Nunes AT, Li M, Marcovitz M, Lanasa MC, Monk BJ. CALLA: Efficacy and safety of concurrent and adjuvant durvalumab with chemoradiotherapy versus chemoradiotherapy alone in women with locally advanced cervical cancer: a phase III, randomized, double-blind, multicenter study. Int J Gynecol Cancer. 2020 Jul;30(7):1065-1070. doi: 10.1136/ijgc-2019-001135. Epub 2020 May 23. PMID 32447296
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9100C00001&attachmentIdentifier=a290db6a-1ec0-4b2d-a142-1d9d56d6fffc&fileName=D9100C00001-CSR_synopsis_Revised_Redacted_PDFA.pdf&versionIdentifier=
- See also: CSR addendum — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9100C00001&attachmentIdentifier=aa6dc71f-9108-4682-ba4e-39a3ef218fde&fileName=d9100c00001-CSR_addendum.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab + SoC CCRT: Durvalumab 1500mg IV infusion every 4 weeks plus Standard of Care (SoC) concurrent chemoradiotherapy (CCRT) (chemotherapy for 5 weeks plus external beam radiotherapy and brachytherapy)
- Placebo + SoC CCRT: Placebo IV infusion every 4 weeks plus Standard of Care (SoC) concurrent chemoradiotherapy (CCRT) (chemotherapy for 5 weeks plus external beam radiotherapy and brachytherapy)
Period: Overall Study
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Started | 385 | 385
Completed | 268 | 249
Not Completed | 117 | 136
Not completed — Death | 90 | 111
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 19 | 16
Not completed — No longer eligible due to additional cancer diagnosis | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT | Total
Number analyzed (Participants) | 385 | 385 | 770
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.6 (11.74) | 48.8 (11.67) | 49.2 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 385 | 770
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 130 | 125 | 255
  Black or African American | 10 | 12 | 22
  Asian | 152 | 148 | 300
  American Indian or Alaska Native | 47 | 56 | 103
  Other | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on the Investigator Assessment According to RECIST 1.1 or Histopathologic Confirmation of Local Tumour Progression
Description: PFS defined as time from date of randomisation until date of tumour progression or death by any cause, regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression
Time Frame: Tumor assessments start 20 weeks after randomisation then every 12 weeks up to 164 weeks, then every 24 weeks until date of RECIST1.1 defined radiological progression. Assessed up to date of DCO (20-Jan-2022) to a maximum of 32.6 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Durvalumab + SoC CCRT vs Placebo + SoC CCRT; Test type: Superiority; p = 0.174, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.65 to 1.08]

2. Secondary Outcome: Progression-free Survival (PFS) Based on the Investigator Assessment According to RECIST 1.1 or Histopathologic Confirmation of Local Tumour Progression, PD-L1 Expression >= 1%
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PD-L1 Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [26.9 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Durvalumab + SoC CCRT vs Placebo + SoC CCRT; Test type: Superiority; p = 0.203, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.10]

3. Secondary Outcome: Overall Survival (Count)
Description: Number of Participants with Overall Survival (OS) where OS was defined as the time from the date of randomisation until death by any cause
Time Frame: Time from date of randomisation until date of death by any cause, assessed up to the data cut-off date (3rd July 2023), assessed up to a maximum of 51.7 months
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Participants
  Died | 91 | 112
  Censored (includes subjects who withdrew consent and subjects who were lost to follow up) | 294 | 273

4. Secondary Outcome: Overall Survival (Duration)
Description: Time from the date of randomisation until death by any cause
Time Frame: as for outcome 3
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Durvalumab + SoC CCRT vs Placebo + SoC CCRT; Test type: Superiority; p = 0.091, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.60 to 1.04]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Percentage of evaluable patients with an Investigator-assessed visit response of complete response (CR) or partial response (PR). CR defined as disappearance of all target and non-target lesions and no new lesions. PR defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Percentage of Participants | 82.6 | 80.5
Statistical Analysis 1: Comparison: Durvalumab + SoC CCRT vs Placebo + SoC CCRT; Test type: Superiority; p = 0.465, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.794 to 1.657]

6. Secondary Outcome: Complete Response Rate
Description: Percentage of evaluable patients with an overall visit response of Complete Response (disappearance of all target and non-target lesions)
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Percentage of Participants | 42.9 | 40.3
Statistical Analysis 1: Comparison: Durvalumab + SoC CCRT vs Placebo + SoC CCRT; Test type: Superiority; p = 0.469, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.833 to 1.487]

7. Secondary Outcome: Duration of Response (DoR) in Patients With Complete Response (CR)
Description: Time from date of first documented CR until date of documented progression or death in the absence of progression. For patients who did not progress their DoR was their Progression-free survival censoring time
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Durvalumab + SoC CCRT | Placebo + SoC CCRT
Number analyzed (Participants) | 385 | 385
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events

ADVERSE EVENTS:
Time Frame: From the time of signature of informed consent throughout the treatment period (median duration of 656 and 532 days for durvalumab and placebo respectively) up to and including the 90-day safety follow-up period following the last dose of study treatment, up to a maximum of 53 months (Data cut-off date of 03Jul2023)
Description: There were 385 subjects randomised to each of Durva + SoC CCRT and Placebo + SoC CCRT respectively (Full Analysis Set), however 1 of the subjects allocated to Placebo + SoC CCRT did not receive treatment (resulting in 384 in the Safety Analysis Set). Hence, for Placebo + SoC CCRT, the Total number at risk for all-cause mortality = 385 while the Total # at Risk by any Serious Adverse Event = 384 and the Total # at Risk by any Other Adverse Event = 384
Groups:
- Durva + SoC CCRT; Placebo + SoC CCRT: Description (Arm-group)
Arm/Group | Durva + SoC CCRT | Placebo + SoC CCRT
All-Cause Mortality (participants affected / at risk) | 91/385 | 112/385
Serious Adverse Events (participants affected / at risk) | 113/385 | 90/384
Other Adverse Events (participants affected / at risk) | 373/385 | 368/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva + SoC CCRT (N=385) | Placebo + SoC CCRT (N=384)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram q wave abnormal (Investigations) | 0 (0) | 1 (1)
Full blood count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 3 (3) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 3 (3)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (5) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 1 (1) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 7 (8) | 5 (5)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 20 (20) | 20 (20)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (2) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (2)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 16 (19) | 11 (15)
Uterine infection (Infections and infestations) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva + SoC CCRT (N=385) | Placebo + SoC CCRT (N=384)
Aspartate aminotransferase increased (Investigations) | 34 (56) | 30 (38)
Blood alkaline phosphatase increased (Investigations) | 21 (30) | 13 (17)
Blood creatinine increased (Investigations) | 31 (48) | 23 (30)
Gamma-glutamyltransferase increased (Investigations) | 30 (41) | 28 (37)
Lymphocyte count decreased (Investigations) | 18 (29) | 34 (47)
Neutrophil count decreased (Investigations) | 74 (216) | 85 (221)
Platelet count decreased (Investigations) | 48 (81) | 62 (107)
Thrombocytopenia (Blood and lymphatic system disorders) | 38 (46) | 28 (38)
Weight decreased (Investigations) | 43 (46) | 42 (53)
White blood cell count decreased (Investigations) | 71 (296) | 85 (340)
Decreased appetite (Metabolism and nutrition disorders) | 89 (103) | 64 (74)
Hyperglycaemia (Metabolism and nutrition disorders) | 26 (28) | 19 (23)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 24 (32) | 25 (34)
Hypokalaemia (Metabolism and nutrition disorders) | 44 (63) | 46 (74)
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 (52) | 38 (61)
Hyponatraemia (Metabolism and nutrition disorders) | 29 (40) | 23 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (51) | 42 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (47) | 43 (45)
Myalgia (Musculoskeletal and connective tissue disorders) | 26 (29) | 14 (18)
Dizziness (Nervous system disorders) | 19 (24) | 20 (25)
Headache (Nervous system disorders) | 42 (55) | 43 (51)
Insomnia (Psychiatric disorders) | 41 (47) | 33 (34)
Dysuria (Renal and urinary disorders) | 61 (74) | 70 (80)
Hyperthyroidism (Endocrine disorders) | 26 (27) | 12 (13)
Pelvic pain (Reproductive system and breast disorders) | 40 (48) | 37 (41)
Vaginal discharge (Reproductive system and breast disorders) | 30 (37) | 28 (31)
Vaginal haemorrhage (Reproductive system and breast disorders) | 24 (28) | 29 (33)
Hypothyroidism (Endocrine disorders) | 60 (68) | 21 (21)
Hot flush (Vascular disorders) | 28 (31) | 21 (24)
Hypertension (Vascular disorders) | 16 (25) | 24 (31)
Abdominal distension (Gastrointestinal disorders) | 20 (21) | 11 (13)
Anaemia (Blood and lymphatic system disorders) | 209 (315) | 200 (322)
Abdominal pain (Gastrointestinal disorders) | 50 (71) | 54 (68)
Abdominal pain upper (Gastrointestinal disorders) | 30 (31) | 20 (23)
Constipation (Gastrointestinal disorders) | 97 (119) | 87 (106)
Diarrhoea (Gastrointestinal disorders) | 177 (257) | 190 (289)
Haemorrhoids (Gastrointestinal disorders) | 14 (14) | 23 (24)
Nausea (Gastrointestinal disorders) | 213 (289) | 202 (293)
Vomiting (Gastrointestinal disorders) | 105 (194) | 107 (202)
Asthenia (General disorders) | 34 (45) | 35 (43)
Fatigue (General disorders) | 52 (55) | 70 (79)
Pyrexia (General disorders) | 35 (51) | 32 (37)
Leukopenia (Blood and lymphatic system disorders) | 59 (100) | 58 (120)
Covid-19 (Infections and infestations) | 29 (29) | 40 (46)
Cystitis (Infections and infestations) | 25 (28) | 19 (21)
Lymphopenia (Blood and lymphatic system disorders) | 39 (59) | 29 (51)
Herpes zoster (Infections and infestations) | 22 (24) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 26 (27) | 14 (19)
Urinary tract infection (Infections and infestations) | 90 (123) | 92 (124)
Neutropenia (Blood and lymphatic system disorders) | 74 (120) | 55 (100)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 20 (21) | 10 (10)
Radiation proctitis (Injury, poisoning and procedural complications) | 25 (27) | 26 (26)
Radiation skin injury (Injury, poisoning and procedural complications) | 17 (18) | 27 (27)
Alanine aminotransferase increased (Investigations) | 43 (64) | 37 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03830866/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT03830866/SAP_002.pdf